CLINICAL TRIAL: NCT05364905
Title: Patients Characteristics, Treatment Pattern & Outcomes of Patients With Advanced, Recurrent or Metastatic Endometrial Carcinoma: A Retrospective Study
Brief Title: Patients Characteristics, Treatment Pattern & Outcomes of Patients With Advanced, Recurrent or Metastatic Endometrial Carcinoma
Acronym: ENDOVIE
Status: Completed | Type: Observational
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GINECO-EN106
Record Dates: First submitted 2022-04-29; First posted 2022-05-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Oncology; Endometrial Cancer; Advanced Cancer; Recurrent Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasms; Endometrial Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients in first line treatment (first chemotherapy for advanced, recurrent or metastatic endometrial cancer) in 2019
  Interventions: Drug: Chemotherapy
- Cohort 2: Patients in second line treatment (after one prior systemic chemotherapy) in 2019
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Patients with confirmed advanced, recurrent or metastatic endometrial cancer, treated by chemotherapy in real life-setting, between 1st January 2019 to 31rd December March 2019, in first or second line of chemotherapy.

SUMMARY:
This is a national observational retrospective multi-site chart review study of patients with advanced, recurrent or metastatic endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women ≥ 18 years at index date.
2. Documented diagnosis of advanced recurrent or metastatic endometrial cancer not eligible to primary complete surgery. Patients with interval surgery after primary CT may be eligible.
3. Index date should represent at least the first* or second line** chemotherapy systemic treatment and occur between, 1, January 2019 and 31, December 2019.
4. do not express refusal to her personal data processing or did not express her refusal for deceased patients.

Exclusion Criteria:

1. No clinical records for tumor imaging or administration of anti-cancer therapy.
2. Patients with active malignancy other than EC cancer which contribute significantly to the clinical impairment of the patient during the study period, according to investigator opinion.
3. Patients lost to follow-up, defined as patients whose last follow-up information occurs less than two years after index date (unless the patient is deceased).
4. Patient did not receive chemotherapy systemic treatment.
5. Patient undergo treatment by pembrolizumab or another immunotherapy in first line (cohort 1) or second line (cohort 2) during the eligibity (inclusion) period.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population musy respect all the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Clinical, biological and treatment characteristics | up to 3 years
  Description of the data

SECONDARY OUTCOMES:
Progession Free Survival real world (rwPFS) | through study completion, an average of 1 year
  From the date of initiation of the treatment in the corresponding line to the date of progression or death
Overall Survival (OS) | through study completion, an average of 1 year
  From the date of initiation of the treatment in the corresponding line to the date of death

CONTACTS AND LOCATIONS:
Locations (30):
- France (30):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Sainte-Catherine Institut du Cancer Avignon-Provence, Avignon
  - CHRU Besançon - Hôpital Jean Minjoz, Besançon
  - Guillaume BABIN, Bordeaux
  - Hôpital Morvan CHRU de Brest, Brest
  - Centre d'Oncologie et de Radiothérapie 37, Chambray-lès-Tours
  - Hôpital Louis Mourier, Colombes
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU de Dijon, Dijon
  - Centre Georges François Leclerc, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - ICL - Centre Alexis Vautrin, Nancy
  - ORACLE - Centre d'Oncologie de Gentilly, Nancy
  - Hôpital Privé du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre ONCOGARD - Institut de cancérologie du Gard, Nîmes
  - CHR Orléans, Orléans
  - Institut Curie, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Groupe Hospitalier Diaconesses - Croix Saint-Simon, Paris
  - Centre CARIO - HPCA, Plérin
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - Centre Eugène Marquis, Rennes
  - ICO - Centre René Gauducheau, Saint-Herblain
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - CHU Tours - Hôpital Bretonneau, Tours
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No